CLINICAL TRIAL: NCT06811155
Title: Non-Interventional, Descriptive, Cross-sectional and Unicentric Study to Describe the Clinical Management in Asthmatic Patients Attended in the Influential Area of Hospital Universitario Virgen de la Victoria, Málaga
Brief Title: Non-Interventional Study to Describe the Clinical Management in Asthmatic Patients (NICMA)
Acronym: (NICMA)
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Virgen de la Victoria (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: FIS-ASP-2020-01
Record Dates: First submitted 2020-10-20; First posted 2025-02-06 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: asthma; clinical management; exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is a heterogenic chronic disease that affects more than 300 million people worldwide, which it's characterized by acute symptomatic episodes of varying severity, including intermittently inflammation and narrowing of the airways in the lungs.

The prevalence in Spain it is estimated to be around 5%, according to the European Community Respiratory Survey (ECRHS) and seems to be increased due to a higher rate of asthma diagnosis.

In this condition there's substantial proportion of patients with a poor disease control, which conducts to an important negative impact in their health-related quality of life (HRQoL) and the need to use health care resources.

During the past decades multiple clinical practice guidelines, such as the international Global Initiative for Asthma (GINA) and national guidelines as Guía Española para el Manejo del Asma (GEMA) have been launched with the aim of improving quality of care in patients with asthma and reduce the high public burden associated to this disease. However, several studies have concluded that high proportion of patients remain uncontrolled, being in Spain estimated around 50%, and there's direct evidence of poor adherence to the guideline's recommendations for asthma management.

This evidence raises the need to determine the assistance quality care in asthma population in the influential area of Hospital Universitario Virgen de la Victoria through the assistance quality care indicators established by GEMA guidelines. The aim of this study is to obtain clinical data that allow to assess assistance quality degree in order to find improvement opportunities to achieve a better control of asthmatic patients within this influential area.

DETAILED DESCRIPTION:
A non-Interventional, descriptive, cross-sectional and unicentric study, has been designed and will be conducted in a Spanish hospital of Málaga. The design of the study imposes an only visit to be performed to obtain the patient's signed IC and after signing it (if patient agreed to participate in the study. Except for this study visit, the rest of study will be based on electronic medical chart review of approximately 300 asthma patients belonging the influential area of Hospital Universitario Virgen de la Victoria. This chart review will be performed by the site investigator or collaborators.

The data collection is stated in 6 months, and during this period the investigators will identify and randomly include the patients who meet selection criteria to avoid bias during patient's inclusion. The observational period will be conformed of 12 months, and the patient's data will be collected or documented in an electronic case report form (eCRF), which will automatically create or assign an identification numerical code to every patient the moment it's created in the electronic platform. This system guarantees the anonymization of each patient included in the study as no identifiable information won't be able to be captured.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with written informed consent prior to participation.
2. Patient female or male ≥ 18 years of age
3. Patient with asthma diagnosis more than one year before the study inclusion
4. Clinical data available at least 1 year before the study inclusion in the electronic medical records.

Exclusion Criteria:

1. Patient's participation in any clinical trial during the year prior to the index date for data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in Hospital Virgen de la Victoria, which it's the reference hospital that usually attends the asthma population of its influential area. Only patients that meet the eligibility criteria will be included in the study, and it is planned that a total estimation of 300 patients with asthma diagnose will be included in it. The whole patients will be recruited by the site investigator and collaborators, who will conduct the subject's medical chart review. Before the patient's study inclusion, the investigator team must have been obtained the signed informed consent of each patient recruited and according to ICH GCP and to local legal requirements.
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HU Virgen de la Victoria, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 305 patients were screened for being included in the study. Of them, 17 patients did not meet all the eligibility criteria, with a final sample size of 288 patients
Groups:
- Asthma Patients: A total of 305 patients were screened for being included in the study. Of them, 17 patients did not meet all the eligibility criteria, with a final sample size of 288 patients
Period: Overall Study
Arm/Group | Asthma Patients
Started | 288
Completed | 288
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 305 patients were screened for being included in the study. Of them, 17 patients did not meet all the eligibility criteria, with a final sample size of 288 patients. Demographic and clinical characteristics of the participating patients are shown in
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Age, Categorical [Count of Participants; unit: Participants] — Mean age at the time of the study visit (SD) (years) is 48.59 (14.91)
  Participants
    <=18 years | 0
    Between 18 and 65 years | 236
    >=65 years | 52
Age, Continuous [Mean (Standard Deviation); unit: YEARS] — Mean age at the time of the study visit (SD) (years) 48.59 (14.91)
  YEARS | 48 (14)
Sex: Female, Male [Count of Participants; unit: Participants] — Female gender, n (%) 185 (64.2%)
  Participants
    Female | 185
    Male | 103
Region of Enrollment [Number; unit: participants] — Adult patients diagnosed with asthma and followed-up in the influential area of Virgen de la Victoria University Hospital, referral hospital in Málaga (Spain)
  participants
    Spain | 288
Race (NIH/OMB) [Count of Participants; unit: Participants] — We classify our population into: white, asian and latino or hispanic.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 272
    More than one race | 0
    Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Clinical Management in Asthmatic Patients
Description: Describe the clinical management in asthmatic patients in the influential area of Hospital Universitario Virgen de la Victoria according to the assistance quality indicators established by GEMA guidelines
Time Frame: Data collected for 6 months
Population: The level of compliance was evaluated in the total study population (n=288) for row number 1, 4 and 6.
  For row number 2, we evaluated those patients included in the study with a history of allergic asthma (n=122).
  For row number 3, we evaluated the patients who were smokers at study entry (n=38).
  For row number 5, we evaluated patients with mild, moderate or severe persistent asthma (n=91).
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Participants
  Asthma diagnosis confirmed by spirometry and bronchodilator test | 60
  Sensitization to allergen study in patients with history of suspected allergic asthma: number analyzed (Participants) | 122
  Sensitization to allergen study in patients with history of suspected allergic asthma | 64
  Smoker patients who were advised on the importance of stopping this habit: number analyzed (Participants) | 38
  Smoker patients who were advised on the importance of stopping this habit | 29
  Patients who were included in an educational plan | 41
  Patient who were receiving inhaled glucocorticoids at inclusion date for persistent asthma treatment: number analyzed (Participants) | 91
  Patient who were receiving inhaled glucocorticoids at inclusion date for persistent asthma treatment | 84
  Patients who had an evaluation and documentation of exacerbations | 40

2. Secondary Outcome: Sociodemographic and Clinical Characteristics
Description: To describe the sociodemographic and clinical characteristics of the study population
Time Frame: Data collected for 6 months
Population: We have only described the most prevalent demographic and clinical characteristic from the patients in the study.
Measure: Number; unit: Participants
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Participants
  Female gender | 185
  White ethnicity | 272
  Positive pregnancy status: number analyzed (Participants) | 185
  Positive pregnancy status | 3
  Chronic pulmonary disease comorbidity | 56
  Patient's management in primary care | 269
  Mild intermittent asthma severity degree according to GEMA guidelines | 197
  Step 1 asthma therapeutic level according to GEMA stepwise therapy | 178

3. Secondary Outcome: Treatment Patterns.
Description: To describe the treatment patterns (maintenance treatment, reliever treatment, type of treatment)
Time Frame: Data collected for 6 months
Population: We have described the treatments patterns from all the patients in the study.
Measure: Number; unit: Participants
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Participants
  Short-acting β2 agonist (SABA) | 76
  long-acting muscarinic antagonist (LAMA) | 14
  Inhaled glucocorticoid (GCI) | 153
  leukotriene receptor antagonist (LTRA) | 25
  Long-acting β agonist (LABA) + Inhaled glucocorticoid (GCI) | 139
  Biologic | 6
  Inmunomodulator | 5
  Oral corticosteroids (OCS) | 35
  Other | 12

4. Secondary Outcome: Level of Disease Control
Description: To describe the disease control level in the study population
Time Frame: Data collected for 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Participants
  ACT score ≥20 (well-controlled asthma) | 158
  ACT score <20 (uncontrolled asthma) | 130

5. Secondary Outcome: Use of Health Resources
Description: To describe the use of health resources (emergency visit, Primary care visits, specialist visits)
Time Frame: Data collected for 6 months
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Visits
  Mean number of emergencies visits due to asthma | 0.07 (0.32)
  Mean number of unscheduled primary care visits due to asthma | 0.13 (0.39)
  Mean number of scheduled primary care visits | 0.12 (0.55)
  Mean number of unexpected primary care visits | 0.13 (0.39)
  Mean number of allergology visits | 0.19 (0.77)
  Mean number of pneumology visits | 0.12 (0.42)

6. Secondary Outcome: Number of Patients With SABA Discontinuation
Description: To describe the number of patients with SABA discontinuation
Time Frame: Data collected for 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Patients
Number analyzed (Participants) | 288
Participants | 28

ADVERSE EVENTS:
Time Frame: Data collected for 6 months
Description: no adverse events
Groups:
- Population: Population Description
Arm/Group | Population
All-Cause Mortality (participants affected / at risk) | 0/288
Serious Adverse Events (participants affected / at risk) | 0/288
Other Adverse Events (participants affected / at risk) | 0/288

LIMITATIONS AND CAVEATS:
The limitations of the study are linked to the retrospective design. The number of spirometry tests used to diagnose asthma may be underestimated. The spirometry tests used for diagnosis were not included in the database. In addition, other variables retrospectively collected from the medical charts may not be routinely recorded or inconsistently recorded by the clinicians (eg, inaccurate filling of the medical records).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT06811155/Prot_SAP_ICF_000.pdf